CLINICAL TRIAL: NCT05330338
Title: Genetics of Ventriculo-arterial Discordance: Towards a PRECIsion Medicine in PEDiatric Cardiology
Brief Title: Genetics of Ventriculo-arterial Discordance
Acronym: PreciPed
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Inserm UMR1087, CNRS UMR6291 (Unknown); Clinique des Données, CIC 1413, CHU Nantes (Unknown); CIC-FEA, CIC 1413, CHU Nantes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC21_0555
Record Dates: First submitted 2022-03-22; First posted 2022-04-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital heart disease; Ventriculo-arterial discordance; Transposition of the great arteries; Transposition congenitally corrected of the great arteries; Genetic; Whole genome sequencing
MeSH Terms: conditions — Heart Defects, Congenital; Transposition of Great Vessels; Congenitally Corrected Transposition of the Great Arteries

STUDY DESIGN:
Intervention Model Description: 900 participants (300 trio families)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Congenital heart disease (Other)
  Interventions: Biological: Genetic analyses: whole genome sequencing

INTERVENTIONS:
Biological: Genetic analyses: whole genome sequencing — Identification of de novo genetic variants using a whole genome sequencing (WGS) approach in the context of familial trios analysis

SUMMARY:
Number of centres planned : 16 centres in France

Type of study / Study design : Research Involving the Human Person category 2.

Multicentric. Prospective

Planning of the study : Total duration: 57,5 months. Recruitment period: 33.5 months. Follow-up time per patients : 2 years

Expected number of cases : The study will involve a maximum of 900 individuals, from 16 centers in France300 family trios (consisting of 150 index cases and their 2 parents, healthy volunteers, N= 450 individuals)

- In the event of unavailability, refusal, non-compliance with an inclusion or exclusion criterion concerning one of the biological parents, only the index case (patient) will be included in the study without his or her parents.

The 300 index cases with ventriculo-arterial discordance will be divided into two groups: 100 double discordance cases and 200 large-vessel transpositions.

These group inclusion targets are theoretical. If the proportion of patients available for inclusion turns out to be higher than expected for one of the groups, the targets may be adjusted, while maintaining a maximum of 300 cases included (corresponding to 900 subjects if all trios are complete).

Patients and their parents will be informed of the study by their referring cardiologist, and their written consent will be obtained.

Translated with DeepL.com (free version)

Treatment, procedure, combination of procedures under consideration :

* Blood samples for genetic analyses collected at the inclusion visit for patients and parents in case of trio families

Schedule of different visits and examinations :

Inclusion visit:

* Collection of demographic, clinical data from the index case and parents
* DNA sampling for genetic research (biocollection) of the index case or family trio
* Completion of the quality of life questionnaire

Annual visit with a 2 years follow-up:

* Retrieval of data from the index case
* Completion of the quality of life questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients with transposition of the great arteries or transposition congenitally corrected of the great arteries with healthy parents and no family history of congenital heart disease (familial trio)
* Or patients with transposition of the great arteries or transposition congenitally corrected of the great arteries with or without a history of congenital heart disease (familial form or sporadic case)
* Affiliated or beneficiaries of a social security scheme or similar
* After obtaining oral consent from patients and/or parents if applicable

Parents (for family trios) :

- Biological parents of the child included in the PRECIPED study

Exclusion Criteria:

* Patients with transposition of the great arteries or transposition congenitally corrected of the great arteries with hypoplastic ventricle or atrioventricular and/or ventriculoarterial valve atresia
* Patient with an identified malformation syndrome
* Patients under guardianship/curatorship
* Patients with State Medical Aid
* Refusal of consent by the patient and/or one of the two parents

Ages: 1 Minute to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Identification new genes/variants involved in congenital heart disease with transposition congenitally corrected of the great arteries, based on whole genome sequencing of familial trios. | 24 months
  Identification of de novo genetic variants using a whole genome sequencing (WGS) approach in the context of familial trios analysis

SECONDARY OUTCOMES:
Evaluation the diagnostic contribution of parental cardiovascular screening in case of ventriculo-arterial discordance (transposition of the great arteries, transposition congenitally corrected of the great arteries) in the index case. | 24 months
  Evolution of diagnostic performance for congenital heart disease in relatives of the index case with ventriculo-arterial discordance following the introduction of parental screening.
Identification new familial forms of ventriculo-arterial discordance. | 24 months
  Identification of genotype/phenotype relationships by studying associations between clinical features and identified genetic variants.
Identification epigenetic modifications by analysis of the epigenome of sporadic forms when genome sequencing is not contributory. | 24 months
  Detection of epigenetic modifications.
Identification allelic variants associated with prognosis and/or response to treatment, with the aim of eventually developing a precision medicine programme in paediatric cardiology | 2 years
  Identification of genotype/phenotype relationships in relation to prognosis and/or response to treatment
Assessing the quality of life of patients with ventriculo-arterial discordance as well as their parents | 2 years
  To document quality of life longitudinally in this patient population using Pediatric Quality of Life InventoryTM (scale from 0 to 4 ; 4 being the worst outcome)
Assessing the quality of life of patients with ventriculo-arterial discordance as well as their parents | 2 years
  To document quality of life longitudinally in this patient population using The Short Form (36) Health Survey (scale from 1 to 6 ; 6 being the worst outcome)

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU Marseille, Marseille, Bouches-du-Rhône
  - CHU Rennes, Rennes, Brittany Region
  - CHU Bordeaux, Bordeaux, Gironde
  - CHU Toulouse, Toulouse, Haute-Garonne
  - CHU de Lille, Lille, Hauts-de-France
  - Groupe Hospitalier St Joseph - Hôpital Marie Lannelongue, Le Plessis-Robinson, Hauts-de-Seine
  - CHU Nantes, Nantes, Loire-Atlantique
  - Hôpital Nord Laennec, Saint-Herblain, Loire-Atlantique
  - CHU Angers, Angers, Maine-et-Loire
  - CHU Nancy, Nancy, Meurthe-et-Moselle
  - Intercard Lille, Lille, Nord
  - CHU de Caen, Caen, Normandy
  - Hôpital Européen Georges Pompidou, Paris, Paris
  - CHU Lyon, Lyon, Rhône
  - CHU Rouen, Rouen, Seine-Maritime
  - CHU Tours, Tours, Val de Loire

IPD SHARING:
Plan to Share IPD: No